CLINICAL TRIAL: NCT05262530
Title: First-in-human, Open-label, Multicenter, Phase I/IIa, Dose Escalation Trial With Expansion Cohorts to Evaluate Safety and Preliminary Efficacy of BNT142 in Patients With CLDN6-positive Advanced Solid Tumors
Brief Title: Safety and Preliminary Efficacy Trial of BNT142 in Patients With CLDN6-positive Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNT142-01; 2021-005481-18 (EudraCT Number); 2024-512639-58-00 (EU CTIS Number)
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
Keywords: CLDN6-positive solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BNT142 (Experimental)
  Interventions: Biological: BNT142

INTERVENTIONS:
Biological: BNT142 — Intravenous bolus/infusion

SUMMARY:
This study is an open-label, multicenter, Phase I/IIa, dose escalation, safety, and pharmacokinetics (PK) study of BNT142 followed by expansion cohorts in patients with Claudin 6 (CLDN6)-positive advanced tumors.

DETAILED DESCRIPTION:
Part 1 (Dose escalation) of this study is a first-in-human (FIH), open-label, dose escalation safety and PK study of BNT142 in patients with advanced/metastatic CLDN6-positive solid tumors.

Part 2 (Expansion) will be a Phase IIa proof-of-concept study in up to three expansion cohorts of CLDN6 positive advanced/metastatic ovarian cancer, non-small cell lung cancer (NSCLC) of non-squamous type, and testicular cancer patients who have progressed on or after last prior treatment.

ELIGIBILITY:
Key Inclusion Criteria:

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

For Part 1 and 2:

* Histological or cytological documentation of a malignant solid tumor (via a pathology report) that is metastatic or unresectable.
* CLDN6-positive tumor sample as assessed by central laboratory testing using a validated immunohistochemistry assay in formalin-fixed paraffin-embedded neoplastic tissues or alternatively from fresh tissue if archival tissue is unavailable. If archival tissue samples from several points of time are available, the most recent one is preferred.
* Measurable disease per RECIST 1.1 (measurable per RECIST 1.1 or evaluable per GCIG criteria for ovarian tumors).

For Part 1 (Dose escalation):

* Patients with advanced/metastatic ovarian (including fallopian tube and peritoneal), non-squamous NSCLC, endometrial, or testicular cancer, for whom there is no available standard therapy likely to confer clinical benefit, or the patient is not a candidate for such available therapy, or patients with not otherwise specified tumors (as confirmed by histological diagnosis), rare tumors (defined as those occurring in <15 out of 100,000 people each year as per National Cancer Institute guidelines) and cancers of unknown primary, not included in the pre-defined eligible tumor types (the last three upon approval by the medical monitor). Patients must have received all available standard therapies, including targeted therapies based on mutation status (per guidelines from the United States Food and Drug Administration [FDA], American Society of Clinical Oncology, European Society for Medical Oncology or local guidelines used at the site), and failed at least first line standard of care therapy prior to enrollment.

Key Exclusion Criteria:

* Chemotherapy, or molecularly-targeted agents within 3 weeks or 5 half-lives (whichever is longer) of the start of study treatment; immunotherapy/monoclonal antibodies within 3 weeks of the start of study treatment; nitrosoureas, antibody-drug conjugates, or radioactive isotopes within 6 weeks of the start of study treatment.
* Radiotherapy in the last 6 weeks prior to the first dose of BNT142 (excluding brain radiotherapy for which 3 weeks prior to the first dose of BNT142 is allowed). Previously irradiated tumor lesions cannot be considered as target lesions or non-target lesions in this study.
* Concurrent systemic (oral or intravenous [IV]) steroid therapy >10 mg prednisone daily or its equivalent for an underlying condition apart from physiologic corticosteroid replacement therapy.
* Major surgery within 4 weeks before the first dose of BNT142.
* Ongoing or active infection requiring IV treatment with anti-infective therapy that has been administered less than 2 weeks prior to the first dose of BNT142.
* Prior treatment with a CLDN6 targeting therapy.
* Side effects of any prior therapy or procedures for any medical condition not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events v.5 Grade ≤1, except for anorexia, fatigue, hyperthyroidism, hypothyroidism, and peripheral neuropathy, which must have recovered to Grade ≤2. Alopecia of any grade is allowed.
* Current evidence of new or growing brain or leptomeningeal metastases during screening. Patients with known brain metastases may be eligible if they:
* Had radiotherapy, surgery or stereotactic surgery for the brain metastases;
* Have no neurological symptoms (excluding Grade ≤2 neuropathy);
* Have stable brain metastasis on the computer tomography (CT) or magnetic resonance imaging (MRI) scan within 4 weeks before signing the informed consent form; and
* Are not undergoing acute corticosteroid therapy or steroid taper.
* Notes: Patients with central nervous system symptoms should undergo a CT scan or MRI of the brain to exclude new or progressive brain metastases. Spinal bone metastases are allowed, unless imminent fracture with cord compression is anticipated.
* Pregnant or breastfeeding or planning to get pregnant within 6 months of the last dose of BNT142.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events (TEAEs) including Grade ≥3, serious, or fatal TEAEs by causal relationship to study treatment | From first dose to 60 days after the last dose of BNT142
Occurrence of dose reductions and discontinuation of BNT142 due to TEAEs | From first dose to 60 days after the last dose of BNT142
Part 1: Occurrence of dose-limiting toxicities (DLTs) during the DLT evaluation period in the dose escalation | Assessed during the DLT period, i.e., up to 5 weeks after first dose of BNT142
Part 2: Objective response rate (ORR) | Up to 36 months after last patient last dose
  ORR is defined as the proportion of patients in whom a confirmed complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, and per Gynecological Cancer Intergroup (GCIG) criteria incorporating RECIST 1.1 and cancer antigen (CA)-125 for the ovarian cancer population is the best overall response.

SECONDARY OUTCOMES:
Part 1: PK parameter: Area under the concentration-time curve in the dosing interval (AUC) | Pre-dose until 60 days after last dose
Part 1: PK parameter: Clearance (CL) | Pre-dose until 60 days after last dose
Part 1: PK parameter: Volume of distribution (Vd) | Pre-dose until 60 days after last dose
Part 1: PK parameter: Maximum observed concentration (Cmax) | Pre-dose until 60 days after last dose
Part 1: PK parameter: Time to maximum observed concentration (Tmax) | Pre-dose until 60 days after last dose
Part 1: PK parameter: Concentration prior to next dose (Ctrough) | Pre-dose until 60 days after last dose
Part 1: PK parameter: Minimum observed concentration (Cmin) | Pre-dose until 60 days after last dose
Part 1: PK parameter: Elimination half-life (t½) | Pre-dose until 60 days after last dose
Part 1: ORR | Up to 36 months after last patient last dose
  ORR (Part 1 only) is defined as the proportion of patients in whom a confirmed CR or PR, per RECIST 1.1, is the best overall response.
Disease control rate (DCR) | Up to 36 months after last patient last dose
  DCR is defined as the proportion of patients in whom a CR or PR or stable disease (SD) (per RECIST 1.1 [and per GCIG criteria for ovarian cancer patients], SD assessed at least 6 weeks after first dose) as best overall response.
Duration of response (DOR) | Up to 36 months after last patient last dose
  DOR is defined as the time from first objective response (CR or PR per RECIST 1.1) to first occurrence of objective tumor progression (progressive disease per RECIST 1.1) or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (18):
- United States (6):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START) - San Antonio, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- National University Cancer Institute - National University Hospital, Singapore, Singapore
- Spain (7):
  - HM Nou Delfos General Hospital, Barcelona
  - Hospital Universitario Vall D'Hebron, Barcelona
  - MD Anderson Cancer Center, Madrid
  - START Madrid-FJD Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre - Centro de Actividades Ambulatorias, Madrid
  - START Madrid CIOCC Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria Campus Universitario de Teatinos, Málaga
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Hammersmith Hospital, Imperial College School Of Medicine - Imperial College Healthcare NHS Trust, London
  - Churchill Hospital - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stadler CR, Ellinghaus U, Fischer L, Bahr-Mahmud H, Rao M, Lindemann C, Chaturvedi A, Scharf C, Biermann I, Hebich B, Malz A, Beresin G, Falck G, Hacker A, Houben A, Erdeljan M, Wolf K, Kullmann M, Chang P, Tureci O, Sahin U. Preclinical efficacy and pharmacokinetics of an RNA-encoded T cell-engaging bispecific antibody targeting human claudin 6. Sci Transl Med. 2024 May 22;16(748):eadl2720. doi: 10.1126/scitranslmed.adl2720. Epub 2024 May 22. PMID 38776391
- [Derived] Simon AG, Lyu SI, Laible M, Woll S, Tureci O, Sahin U, Alakus H, Fahrig L, Zander T, Buettner R, Bruns CJ, Schroeder W, Gebauer F, Quaas A. The tight junction protein claudin 6 is a potential target for patient-individualized treatment in esophageal and gastric adenocarcinoma and is associated with poor prognosis. J Transl Med. 2023 Aug 17;21(1):552. doi: 10.1186/s12967-023-04433-8. PMID 37592303